CLINICAL TRIAL: NCT01557738
Title: Acute and Long-term Effects of Dietary Flavanols on Local Control of Skeletal Muscle Blood Flow During Exercise in Young and Old Humans
Brief Title: Role of Flavanols in Exercise and Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Robert M. Brothers, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012-02-0114
Record Dates: First submitted 2012-03-08; First posted 2012-03-19 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-05

CONDITIONS: Aging
Keywords: Exercise; Blood Flow; Nitric Oxide; Aging; Antioxidant; Flavanol; Young (18-30 yrs); Aging (60 - 80 yrs)
MeSH Terms: conditions — Motor Activity | interventions — Time

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Acute effects of flavanol consumption (Experimental): The outcome measurements will be made on all study participants before and 2 hours after consumption of the high flavanol beverage.
  Interventions: Dietary Supplement: High Flavanol Trial
- Low Flavanol Trial; acute effects (Placebo Comparator): Once again, the outcome measurements will be made on all study participants before and 2 hours after consumption of the low flavanol beverage.
  Interventions: Dietary Supplement: Low Flavanol Trial
- Long-term effects of flavanol consumption (Experimental): Only those study participants over 60 years of age will continue with this arm of the trial. The same outcome measures will be performed following 4 weeks of daily consumption of a high flavanol beverage.
  Interventions: Dietary Supplement: High Flavanol Trial; long-term
- Low Flavanol Trial; long-term effects (Placebo Comparator): Only those study participants over 60 years of age will continue with this arm of the trial. The same outcome measures will be performed following 4 weeks of daily consumption of a low flavanol beverage.
  Interventions: Dietary Supplement: Low Flavanol Trial; long-term effects

INTERVENTIONS:
Dietary Supplement: High Flavanol Trial — The experimental trial (high flavanol content) will involve the consumption of a beverage containing about 1000mg of cocoa flavanols.
  Arms: Acute effects of flavanol consumption
Dietary Supplement: Low Flavanol Trial — The placebo trial (low flavanol content) will involve the consumption of a beverage containing 75 mg of cocoa flavanols.
  Arms: Low Flavanol Trial; acute effects
Dietary Supplement: High Flavanol Trial; long-term — The experimental trial (high flavanol content) will involve the daily consumption of a beverage containing about 1000mg of cocoa flavanols for 4 weeks. Subjects will be provided with 28 packets of the beverage to take home with them.
  Arms: Long-term effects of flavanol consumption
Dietary Supplement: Low Flavanol Trial; long-term effects — The placebo trial (low flavanol content) will involve the daily consumption of a beverage containing 75 mg of cocoa flavanols for 4 weeks. Subjects will be provided with 28 packets to take home with them.
  Arms: Low Flavanol Trial; long-term effects

SUMMARY:
It has well known that diets rich in fruits, vegetables and cocoa products are associated with positive health benefits and these positive effects have been shown to be due to compounds they contain called flavanols. Flavanols have been shown to exert their positive effects by indirectly increasing nitric oxide (NO) bioavailability. NO is a potent vasodilator that is believed to play a role in increasing blood flow to active muscle during exercise. This regulatory process is impaired with healthy aging. The underlying premise to this study is that if NO bioavailability can be increased following flavanol ingestion, will there be a restoration of blood flow during exercise in older individuals? Accordingly, the first part of this research project will compare the acute vascular effects of flavanol ingestion between a young and old group. The investigators have hypothesized that both groups will show an improvement in blood flow to active muscle during exercise, though the magnitude of the change will be greater in the older group. The second part of this project will look at the effects of 4 weeks of daily flavanol ingestion in the old group. The investigators hypothesize that subjects will demonstrate an improvement in blood flow to active muscle during exercise after the 4 week intervention and that the magnitude of the change will be greater than the acute effects. Findings from this proposal will provide evidence for the efficacy of flavanols to be used (as a simple and safe lifestyle intervention) to reverse or combat impaired blood flow regulation in older individuals.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between 18 - 30 years old
* Males and Females between 60 - 80 years old

Exclusion Criteria:

* cardiovascular and/or microvascular disease
* blood clotting disorder
* pregnant lady
* current smoker (or regularly smoked within last year)
* a history of an adverse reaction to cold
* taking medications known to effect the autonomic nervous system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in femoral blood flow during exercise following flavanol consumption | During knee extension exercise, change from baseline in blood flow 2 hours post flavanol ingestion
  Blood flow regulation to active muscles during knee extension exercise can be assessed by using ultrasound to measure blood flow in the femoral artery. This will be done before and after stimulation of the sympathetic nervous system. A baseline value will be obtained and then the measurement will be performed again 2 hours after flavanol ingestion.

SECONDARY OUTCOMES:
Change in flow-mediated dilation (FMD) following flavanol consumption | Change from baseline in FMD 2 hours post flavanol ingestion
  Flow-mediated dilation is commonly used as an index of nitric oxide bioavailability. Nitric oxide is believed to play a role in blood flow regulation during exercise. A baseline value will be obtained and then the measurement will be performed again 2 hours after flavanol ingestion.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Harrison, M.A., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin: Environmental and Autonomic Physiology Laboratory, Austin, Texas, United States